CLINICAL TRIAL: NCT01488370
Title: A Comparison of the Glidescope® Video Laryngoscope and the Storz DCI® Video Laryngoscope for Endotracheal Intubation in Children Younger Than Two Years of Age
Brief Title: Comparison of 2 Laryngoscopes for Endotracheal Intubation in Children Younger Than 2 Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Elizabeth Ghazal, MD, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 5110244
Record Dates: First submitted 2011-11-01; First posted 2011-12-08 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Endotracheal Intubation
Keywords: breathing tube placement
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glidescope (Active Comparator): A device for endotracheal intubation.
  Interventions: Device: Endotracheal intubation
- Storz (Active Comparator): A device for endotracheal intubation.
  Interventions: Device: Endotracheal intubation
- Standard Laryngoscope (Active Comparator): A device for endotracheal intubation
  Interventions: Device: Endotracheal intubation

INTERVENTIONS:
Device: Endotracheal intubation — Endotracheal intubation
  Other Names: Storz DCI video laryngoscope; Glidescope video laryngoscope

SUMMARY:
This is a prospective randomized clinical study to be performed in pediatric patients under the age of 2 years who are undergoing surgical procedures requiring endotracheal intubation. Time to endotracheal intubation will be compared between patients intubated using a GlideScope® video laryngoscope, those intubated with a Storz DCI® video laryngoscope, and those intubated by standard direct laryngoscopy. The study hypothesis is that the time to endotracheal intubation will be decreased in the Storz DCI® video laryngoscope group when compared to the GlideScope® video laryngoscope group and standard laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients under the age of 2 years undergoing surgeries requiring endotracheal intubation at LLUMC will be eligible for participation in this study

Exclusion Criteria:

* Children with increased pulmonary aspiration risk;
* Prior documentation of difficult endotracheal intubation;
* Those that lack legal representative consent

Max Age: 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2011-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ghazal, MD, Principal Investigator — Loma Linda University Department of Anesthesiology
Locations (2):
- United States (2):
  - Loma Linda University Department of Anesthesiology, Loma Linda, California
  - Loma Linda University Medical Center, Loma Linda, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glidescope | Storz | Standard Laryngoscope
Started | 22 | 23 | 20
Completed | 22 | 22 | 19
Not Completed | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glidescope | Storz | Standard Laryngoscope | Total
Number analyzed (Participants) | 22 | 22 | 19 | 63
Age, Continuous [Median (Full Range); unit: Months] | 7.6 [4.8 to 10.8] | 8.5 [6.3 to 10.5] | 8.1 [5.7 to 13.1] | 8.1 [4.8 to 13.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 6 | 26
  Male | 11 | 13 | 13 | 37
ASA Status I [Count of Participants; unit: Participants] — ASA status was assigned based on standard American Society for Anesthesiologists guidelines, ASA I = healthy. All patients undergoing an anesthetic are assigned and ASA status.
  Participants | 6 | 3 | 4 | 13
ASA Status II [Count of Participants; unit: Participants] — ASA status was assigned based on standard American Society for Anesthesiologists guidelines. ASA II = mild systemic disease. All patients undergoing an anesthetic are assigned and ASA status.
  Participants | 13 | 12 | 9 | 34
ASA Status III [Count of Participants; unit: Participants] — ASA status was assigned based on standard American Society for Anesthesiologists guidelines. ASA III = moderate to severe systemic disease. All patients undergoing an anesthetic are assigned and ASA status.
  Participants | 3 | 5 | 6 | 14
ASA Status IV [Count of Participants; unit: Participants] — ASA status was assigned based on standard American Society for Anesthesiologists guidelines. ASA IV = severe systemic disease that is a constant threat to life. All patients undergoing an anesthetic are assigned and ASA status.
  Participants | 0 | 2 | 0 | 2
Weight [Mean (Full Range); unit: Kg] | 8.2 [7.1 to 9.3] | 8.0 [6.0 to 9.1] | 8.0 [6.9 to 9.2] | 8.0 [6.0 to 9.3]
Percentile Weight for Length [Median (Full Range); unit: Percentile] | 71.9 [49.2 to 84.6] | 58.5 [31.3 to 76.7] | 72.1 [47.6 to 84.0] | 71.9 [31.3 to 84.6]

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Time to Intubation Will Begin at the Time of Mouth Opening and End With the Removal of the Tip of the Laryngoscope Blade From the Patient's Mouth After Successful Endotracheal Intubation.
Time Frame: Less than one day, representing the day of surgery and period of endotracheal intubation during induction of general anesthesia
Population: Time to successful tracheal intubation
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Glidescope | Storz | Standard Laryngoscope
Number analyzed (Participants) | 20 | 21 | 19
Seconds | 30.8 [24.1 to 46.4] | 42.1 [34.0 to 59.0] | 21.5 [17.0 to 34.3]

2. Secondary Outcome: Successful Intubation After One Laryngoscopy Attempt
Description: Other secondary outcome measures will be the use of external laryngeal manipulation to improve glottic view, tissue trauma and type,and method of rescue if initial intubation attempt proves unsuccessful.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Glidescope | Storz | Standard Laryngoscope
Number analyzed (Participants) | 22 | 22 | 19
Participants | 17 | 16 | 16

3. Secondary Outcome: Successful Intubation After Two Laryngoscopy Attempts
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Glidescope | Storz | Standard Laryngoscope
Number analyzed (Participants) | 22 | 22 | 19
Participants | 3 | 5 | 2

4. Secondary Outcome: Successful Intubation After Three Laryngoscopy Attempts
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Glidescope | Storz | Standard Laryngoscope
Number analyzed (Participants) | 22 | 22 | 19
Participants | 1 | 1 | 1

5. Secondary Outcome: Successful Intubation After Four Laryngoscopy Attempts
Time Frame: Through endotracheal intubation during induction of general anesthesia, an average of 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Glidescope | Storz | Standard Laryngoscope
Number analyzed (Participants) | 22 | 22 | 19
Participants | 1 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Glidescope | Storz | Standard Laryngoscope
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/19

LIMITATIONS AND CAVEATS:
Trainees reported more prior intubation experience using DL than the other laryngoscopes, so we were unable to equalize prior clinical experience between DL & other laryngoscopes. Assessment of learning effect limited by intubation types within study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes